CLINICAL TRIAL: NCT06390657
Title: Radiotherapy Treatment Planning Comparison Using SBRT-PATHY (Photons) Versus CARBON-PATHY for Unresectable Bulky Tumors
Acronym: S-C-PATHY
Status: Withdrawn | Type: Observational
Why Stopped: the project was not started.
Sponsor: EBG MedAustron GmbH (Industry)
Collaborators: The Princess Margaret Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: S-C-PATHY-MA-122022
Record Dates: First submitted 2024-03-29; First posted 2024-04-30 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: Particle Radiotherapy; Partial Tumor Irradiation
MeSH Terms: conditions — Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase A: retrospective planning study: Simulation CTs of up to ten patients with bulky (>6cm) tumors will be selected. This will be used for optimization of contouring and planning strategy.
  Interventions: Other: Planning CT, MRI
- Phase B: prospective planning study: Ten patients with bulky tumors (>6cm) recommended to receive RT with CT and MRI planning will be accrued. MRI DCE sequence (20-30mins) will be added if not requested for clinical use. They will be treated with standard clinical plans. Every effort will be made to include equal numbers of patients (2-3) from head and neck, thorax, abdomen and pelvis. Planning images will be used for the purpose of dosimetric comparison between SBRT-PATHY and CARBON-PATHY radiation plans.
  Interventions: Other: Planning CT, MRI

INTERVENTIONS:
Other: Planning CT, MRI — SBRT-PATHY and CARBON-PATHY planning is performed for study purposes only. Patients will be treated according to standard radiotherapy as per institutional policies.
  The planning images (CT, MRI) will be anonymized and used for planning purposes only.

SUMMARY:
This study uses a novel unconventional radiotherapy technique, consisting of high dose PArtial Tumor irradiation targeting exclusively the HYpoxic segment of unresectable bulky tumors delivered either with photons (SBRT-PATHY) or with carbon-ions (CARBON-PATHY) while sparing the peritumoral immune microenvironment (PIM).

DETAILED DESCRIPTION:
This study will be conducted as a two phase study. Phase A is a retrospective study. Up to 10 patients with bulky (>6cm tumors) previous planned with planning CT with IV contrast will be selected for planning and dosimetry comparison. This is performed to optimize the contouring and planning procedures. Phase B is a prospective study. Ten patients with bulky (>6cm tumor) requiring radiotherapy, with planning CT and MR with IV contrast will be accrued. Every effort will be made to include equal numbers of patients (2-3) from head and neck, thorax, abdomen and pelvis. Their images will be used for planning and dosimetry comparison.

Patients will be treated according to clinical plans. The study plans will not be used for treatment. Treatment plans for Photon delivery (SBRT-PATHY) and Carbon delivery (CARBON-PATHY) to deliver 30 Gy in three fractions will be planned to be delivered to the BTV will be performed. SBRT-PATHY plans will be generated at the Princess Margaret Cancer Center (PMCC, Toronto, Canada) while CARBON-PATHY plans will be generated at the MedAustron Center for Particle Therapy and Research (W. Neustadt, Austria).

The objective is to compare the dosimetric profile achievable using SBRT-PATHY (using photons) and CARBON-PATHY (using carbon-ions) for unresectable bulky tumors and surrounding tissues.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (for use their planning CT and MR data for study specific planning)
2. Malignant solid bulky primary or recurrent tumor with diameter of ≥6 cm
3. Age > 18 years
4. Radiation planning CT (with IV contrast) and MRI (with or without IV contrast) is planned

Exclusion Criteria:

1. Patients without bulky lesions,
2. Contraindication to i.v. CT and MRT contrast medium administration, particularly estimated glomerular filtration rate (GFR) less than 45 mL/min/1.73 m².
3. Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control,
4. Any condition that, in the opinion of the investigators, would interfere with treatment planning or interpretation of study results

Note (1): criterion n°4 will be evaluated on the four eyes principle, evaluated by both Principle Investigator and Sub-Investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable bulky tumors (primary or metastatic) recommended to receive external beam radiotherapy, will be recruited from Princess Margaret Cancer Center and Medaustron. Every effort will be made to equal numbers (i.e. 2-3) from head and neck, thorax, abdomen, pelvis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase A: optimization of contouring and planning using PATHY strategy | 18 months (phase A and B combined)
  The objective of phase A is to optimize the target delineation, planning strategy and techniques for SBRT-PATHY at Princess Margaret and CARBON-PATHY at MedAustron.
Phase B: optimal coverage of Bystander tumor volume (BTV) while allowing the maximal radiation-sparing of PIM and regional lymph nodes | 18 months (phase A and B combined)
  a prospective identification of 10 patients who are recommended to receive radiotherapy fulfilling the inclusion criteria. SBRT-PATHY and CARBON-PATHY planning is perfomed for study purposes only. A planning comparison between SBRT-PATHY (using photons) and CARBON-PATHY (using carbon-ions) based on dosimetric consideration achieved for the targeted BTV, non-targeted surrounding NTV (normoxic tumor segment), PIM, regional metastases (i.e. local regional involved nodes and distant metastases located within 15 cm cranial caudal to GTV), regional uninvolved lymph nodes and surrounding organs at risk (OAR) will be performed.

SECONDARY OUTCOMES:
Phase B: Dosimetric-sparing of normoxic tumor volume (NTV) | 18 months (phase A and B combined)
  The normoxic tumor segment (NTV) will be created by subtracting the BTV from the GTV, representing the remaining peripheral tumor segment outside the BTV.
Phase B: Dosimetric-sparing of Organs at risk (OAR) and regional nodes | 18 months (phase A and B combined)
  The OAR will be delineated on MRT images at the level of the treated area. Particularly normal structures involved by or in the close proximity to the tumor such as vessels, nerves, or hollow organs will be contoured. Contours will be checked and refined on the co-registered simulation CT images.
Phase B: Feasibility for dosimetric-sparing of regional/distant metastases as abscopal tumor sites (if present) | 18 months (phase A and B combined)
  Abscopal tumor site(s), corresponding to radiographic evidence of the regional (for ex. lymph nodes) metastases, will be delineated on whichever images that clearly demonstrate their presence, including simulation CT or MRT.

CONTACTS AND LOCATIONS:
Overall Officials: Slavisa Tubin, M.D., Principal Investigator — EBG MedAustron; Rebecca Wong, MBChB, FRCPC, MSc, Prof., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- EBG MedAustron GmbH, Wiener Neustadt, Lower Austria, Austria